CLINICAL TRIAL: NCT01300923
Title: Pilot Study of Acamprosate in Youth With Fragile X Syndrome
Brief Title: Acamprosate in Youth With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1003-26
Record Dates: First submitted 2010-08-25; First posted 2011-02-23 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Fragile X Syndrome; Autism Spectrum Disorders
Keywords: Fragile X Syndrome; Acamprosate
MeSH Terms: conditions — Fragile X Syndrome; Autism Spectrum Disorder | interventions — Acamprosate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acamprosate (Active Comparator): The maximum dose of acamprosate to be used in this study is 1998 mg per day for those subjects weighing greater than 60kg and 1332 mg per day for those less weighing less than 60kg.
  Interventions: Drug: Acamprosate
- Autism Spectrum Disorder (No Intervention): This baseline comparison group will participated in only the psychophysiological and biomarker portion of subject characterization.

INTERVENTIONS:
Drug: Acamprosate
  Other Names: Campral
  Arms: Acamprosate

SUMMARY:
Fragile X syndrome (FXS) is the most common inherited form of developmental disability. FXS is inherited from the carrier parent, most often the mothers. FXS is associated with severe interfering behavioral symptoms which include anxiety related symptoms, attention deficit hyperactivity, and aggressive behaviors. Approximately 25-33% of individuals with FXS also meet criteria for autistic disorder. The hypothesis of this study is that treatment with acamprosate will reduce inattention/hyperactivity, language impairment, irritability, social deficits, and cognitive delay in youth with FXS. The purpose of this study is to investigate the effectiveness and tolerability of acamprosate in youth with Fragile X Syndrome and to assess the potential psychophysiological differences between FXS and autism spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients between the ages of 5 and 17 years.
* Confirmed diagnosis of Fragile X Syndrome based upon genetic testing.
* Stable dosing of all psychotropic medications for at least 2 weeks prior to baseline.
* Subjects with a stable seizure disorder or history of only childhood febrile seizures will be included.
* Clinical Global Impression-Severity Score of 4 (Moderately Ill) or greater.
* Must be in good physical health.
* Subjects of child bearing age of both genders will be required to utilize birth control as applicable.

Exclusion Criteria:

* Diagnosis of schizophrenia, another psychotic disorder, bipolar disorder or alcohol or other substance abuse based on Diagnostic and Statistical Manual Fourth Edition-Text Revised (DSM-IV-TR).
* A significant medical condition such as heart, liver, renal or pulmonary disease or unstable seizure disorder.
* Females with a positive urine pregnancy test
* Creatinine clearance of less than 30.
* Concomitant use of another glutamatergic agent (memantine,riluzole, d-cycloserine, amantadine topiramate, gabapentin, among others.
* Evidence of hypersensitivity to acamprosate or potentially serious adverse effect.
* Subjects who, in the opinion of the investigator, are unsuitable in any other way to participate in this study including being unable to comply with the requirements of the study for any reason.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Erickson, M.D., Principal Investigator — Indiana University School of Medicine - Department of Psychiatry
Locations (1):
- Riley Child and Adolescent Psychiatry Clinic - Riley Hospital for Children, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Erickson CA, Wink LK, Ray B, Early MC, Stiegelmeyer E, Mathieu-Frasier L, Patrick V, Lahiri DK, McDougle CJ. Impact of acamprosate on behavior and brain-derived neurotrophic factor: an open-label study in youth with fragile X syndrome. Psychopharmacology (Berl). 2013 Jul;228(1):75-84. doi: 10.1007/s00213-013-3022-z. Epub 2013 Feb 24. PMID 23436129

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The psychophysiological measures proved non-feasible as subjects could not tolerate the procedures. The paradigms were tried on two subjects in the Autism Spectrum Disorder arm; however, the data that was collected was not usable. Subsequently, neurobiological characterization was halted.
Groups:
- Acamprosate: The maximum dose of acamprosate to be used in this study is 1998 mg per day for those subjects weighing greater than 60kg and 1332 mg per day for those less weighing less than 60kg.
  Acamprosate
- Autism Spectrum Disorder (ADS): This baseline comparison group will participated in only and biomarker portion of subject characterization.
Period: Overall Study
Arm/Group | Acamprosate | Autism Spectrum Disorder (ADS)
Started | 12 | 2
Completed | 12 | 0
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Acamprosate Treatment Group: Twelve subjects received open-label acamprosate, mean final of 1,054 mg/day (range: 666-1,998 mg/day)
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 11.9 [6 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 12
Aberrant Behavior Checklist [Mean (Standard Deviation); unit: units on a scale] — Aberrant Behavior Checklist (ABC) is a 58-item rating scale assessing maladaptive behaviors across 5 original subscales: Irritability(15 items from 0-45), Social Withdrawal(16 items from 0-48), Stereotypy(7 items from 0-21), Hyperactivity(16 items from 0-48), Inappropriate Speech(4 items from 0-12). Also reported is Social Avoidance, a newly developed 4-item subscale (from 0-12) that captures core social avoidance aspects of Fragile X Syndrome. Items on the ABC are rated from 0 (not at all a problem) to 3 (the problem is severe in degree). Higher scores indicate greater maladaptive behaviors.
  units on a scale
    ABC Irritability | 9.9 (7.8)
    ABC Social Withdrawal | 8.8 (5.8)
    ABC Stereotypy | 6.8 (6.8)
    ABC Hyperactivity | 16.8 (9.1)
    ABC Inappropriate Speech | 5.2 (3.5)
    ABC Social Avoidance | 3.3 (2.6)
Clinical Global Impression -Severity [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  units on a scale | 4.25 (0.45)
Children's Yale-Brown Obsessive Compulsive Scale Modified for PDD [Mean (Standard Deviation); unit: units on a scale] — The Children's Yale-Brown Obsessive Compulsive Scales-Modified (CY-BOCS) is a 5-item, semi-structured clinician rating scale modified designed to rate the current severity of repetitive behavior in children and adolescents with PDD. Once the current repetitive behaviors are identified, they are separately rated on 5 items: Time Spent, Interference, Distress, Resistance, and Control. Each of these items is scored on a 5-point scale form 0 (least symptomatic) to 4 (most symptomatic). The CY-BOCS yields a Total Score from 0 to 20 and is sensitive to change.
  units on a scale | 11.1 (2.6)
Social Responsiveness Scale [Mean (Standard Deviation); unit: units on a scale] — The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows: 0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment
  units on a scale | 91.3 (27.4)
ADHD Rating Scale 4th Edition [Mean (Standard Deviation); unit: units on a scale] — The ADHD Rating Scale is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder. The ADHD Rating Scale-IV is completed by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. The total score can range from 0 to 54, with a higher score indicating greater severity.
  units on a scale | 23.6 (10.6)
Peabody Picture Vocabulary Test [Mean (Standard Deviation); unit: units on a scale] — The Peabody Picture Vocabulary Test is one of the most commonly used assessment tests that measure verbal ability in standard American English vocabulary. This test has been nationally standardized using examinees from various age groups, from children to adults. Thus, the raw scores are equated to mental age, using the norms obtained from standardization. The total standard scores range from 40 (worse receptive vocabulary) to 160 (better receptive vocabulary). The scores can also be converted to percentile rank.
  units on a scale | 85.2 (32.0)
Vineland Adaptive Behavior Scales-II (VABS-II) Communication Domain [Mean (Standard Deviation); unit: units on a scale] — The VABS-II is a semi-structured interview designed to assess adaptive functioning in communication, daily living, socialization and motor skills. Recognizing that language is a major area of impairment in the study population, the Communication Domain (99 Items from 0-198), in particular the Expressive Subdomain (54 Items from 0-108) are of interest to this study. Items arranged in a developmental sequence are rated on a 3-point scale. Each item is rated from 0 (never performs the behavior) to 2 (usually performs behavior independently). Higher scores indicate higher adaptive functioning.
  units on a scale
    Communication Domain | 63.4 (10.0)
    Expressive Communication Domain | 69.8 (23.0)
Brain-derived neurotropic factor [Mean (Standard Deviation); unit: pg/mL] — Brain-derived neurotrophic factor (BDNF) is a protein that supports the survival of existing neurons and growth and differentiation of new neurons and synapses.
  pg/mL | 790.4 (1.3050)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression- Severity Scale (CGI-S)
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
units on a scale | 7.0 (8.9)

2. Secondary Outcome: The Aberrant Behavior Checklist (ABC)
Description: The Aberrant Behavior Checklist (ABC) is a 58-item rating scale used to assess maladaptive behaviors across five original subscales: Irritability (15 items from 0-45), Social Withdrawal (16 items from 0-48), Stereotypy (7 items from 0-21), Hyperactivity (16 items from 0-48), Inappropriate Speech (4 items from 0-12). Additionally, Social Avoidance, a newly developed four-item subscale (from 0-12) of the ABC that captures core social avoidance aspects of Fragile X Syndrome is reported. All items on the ABC are rated from 0 (not at all a problem) to 3 (the problem is severe in degree). Higher scores indicate greater maladaptive behaviors. Differences between Baseline and Week 10 are used as an indicator of change.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
units on a scale
  ABC Irritability | 7.0 (8.9)
  ABC Social Withdrawal | 4.1 (6.5)
  ABC Stereotypy | 6.0 (6.3)
  ABC Hyperactivity | 11.0 (8.6)
  ABC Inappropriate Speech | 4.8 (3.4)
  ABC Social Avoidance | 1.6 (2.7)

3. Secondary Outcome: Social Responsiveness Scale
Description: The 65-item SRS is a standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows: 0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
units on a scale | 76.4 (26.8)

4. Secondary Outcome: Children's Yale-Brown Obsessive Compulsive Scale Modified for PDD
Description: The Children's Yale-Brown Obsessive Compulsive Scales-Modified (CY-BOCS) is a 5-item, semi-structured clinician rating scale modified designed to rate the current severity of repetitive behavior in children and adolescents with PDD. Once the current repetitive behaviors are identified, they are separately rated on 5 items: Time Spent, Interference, Distress, Resistance, and Control. Each of these items is scored on a 5-point scale form 0 (least symptomatic) to 4 (most symptomatic). The CY-BOCS yields a Total Score from 0 to 20 and is sensitive to change.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
units on a scale | 9.8 (4.1)

5. Secondary Outcome: ADHD Rating Scale 4th Edition
Description: The ADHD Rating Scale is an 18-item scale directly derived from DSM-IV criteria for Attention Deficit Hyperactivity Disorder. The ADHD Rating Scale-IV is completed by the parent and scored by a clinician. The scale consists of 2 subscales: inattention (9 items) and hyperactivity-impulsivity (9 items). If 3 or more items are skipped, the clinician should use extreme caution in interpreting the scale. The total score can range from 0 to 54, with a higher score indicating greater severity.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
units on a scale | 16.7 (8.0)

6. Secondary Outcome: Vineland Adaptive Behavior Scales-II (VABS-II) Communication Domain
Description: The VABS-II is a semi-structured interview designed to assess adaptive functioning in communication, daily living, socialization and motor skills. Recognizing that language is a major area of impairment in the study population, the Communication Domain (99 Items from 0-198), in particular the Expressive Subdomain (54 Items from 0-108) are of interest in this study. Items arranged in a developmental sequence are rated on a 3-point scale. Each item is scored from 0 (never performs the behavior) to 3 (usually performs the behavior independently). Higher scores indicate higher adaptive functioning. Differences between Baseline and Week 10 are used as an indicator of change.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
units on a scale
  Communication Domain | 66.6 (11.2)
  Expressive Communication | 78.9 (21.2)

7. Secondary Outcome: Peabody Picture Vocabulary
Description: The Peabody Picture Vocabulary Test is one of the most commonly used assessment tests that measure verbal ability in standard American English vocabulary. This test has been nationally standardized using examinees from various age groups, from children to adults. Thus, the raw scores are equated to mental age, using the norms obtained from standardization. The total standard scores range from 40 (worse receptive vocabulary) to 160 (better receptive vocabulary). The scores can also be converted to percentile rank.
Time Frame: Week 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 12
units on a scale | 83.3 (32.0)

8. Secondary Outcome: Brain-derived Neurotrophic Factor (BDNF)
Description: BDNF is a protein that supports the survival of existing neurons and growth and differentiation of new neurons and synapses.
Time Frame: Screen and Week 10
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Acamprosate Treatment Group
Number analyzed (Participants) | 10
pg/mL | 1,007.6 (1,493.2)

ADVERSE EVENTS:
Time Frame: Ten Weeks
Arm/Group | Acamprosate
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acamprosate (N=12)
Irritability (Psychiatric disorders) | 4 (4)
Increased repetitive behavior (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
mild constipation (Gastrointestinal disorders) | 1 (1)
Increased anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Nightmares (Psychiatric disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Psychophysiological measures proved non-feasible as subjects could not tolerate the procedures. The paradigms were tried on 2 subjects in the ADS arm, as data collected was not usable. Subsequently, neurobiological characterization was halted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No